CLINICAL TRIAL: NCT01282333
Title: Phase I Study of Veliparib (ABT-888) in Combination With Cisplatin Plus Gemcitabine in Advanced Biliary, Pancreatic, Urothelial, and Non-small Cell Lung Cancer
Brief Title: Veliparib, Cisplatin, and Gemcitabine Hydrochloride in Treating Patients With Advanced Biliary, Pancreatic, Urothelial, or Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02576; UPCI 10-037; CDR0000693751; PCI-10-037; U01CA099168 (NIH)
Record Dates: First submitted 2011-01-22; First posted 2011-01-25 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Advanced Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer; Metastatic Transitional Cell Cancer of the Renal Pelvis and Ureter; Regional Transitional Cell Cancer of the Renal Pelvis and Ureter; Stage III Bladder Cancer; Stage III Pancreatic Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Bladder Cancer; Stage IV Non-small Cell Lung Cancer; Stage IV Pancreatic Cancer; Transitional Cell Carcinoma of the Bladder; Unresectable Extrahepatic Bile Duct Cancer; Unresectable Gallbladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; veliparib; Cisplatin

ARMS (1):
- Treatment (veliparib, gemcitabine hydrochloride, cisplatin) (Experimental): Patients receive veliparib orally every 12 hours on days 1-12, gemcitabine hydrochloride IV over 30 minutes on days 3 and 10, and cisplatin IV over 60-120 minutes on day 3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with suspected or known germline BRCA mutations may continue to receive single-agent veliparib continuously in the absence of disease progression or unacceptable toxicity. Patients may undergo blood, tumor tissue, and hair follicle sample collection periodically for pharmacokinetic and correlative studies.
  Interventions: Drug: gemcitabine hydrochloride; Drug: veliparib; Other: diagnostic laboratory biomarker analysis; Other: pharmacological study; Drug: cisplatin

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: veliparib — Given orally
  Other Names: ABT-888
Other: diagnostic laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP

SUMMARY:
This phase I clinical trial is studying the side effects and best dose of veliparib and gemcitabine hydrochloride when given with cisplatin in treating patients with advanced biliary, pancreatic, urothelial, or non-small cell lung cancer. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Veliparib may help cisplatin and gemcitabine hydrochloride work better by making tumor cells more sensitive to the drugs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum-tolerated dose of veliparib (ABT-888) (days 1-12 of a 21-day schedule) in combination with cisplatin (day 3) and gemcitabine (days 3, 10) in patients with advanced, previously untreated carcinoma of the bile ducts, gallbladder or pancreas, non-small cell lung cancer, or transitional cell carcinoma of the bladder/urothelial tract.

SECONDARY OBJECTIVES:

I. Describe the dose-limiting toxicity (DLT) and other toxicities associated with veliparib in combination with cisplatin plus gemcitabine as assessed by CTCAE v4.0.

II. Determine the recommended phase 2 dose of veliparib (ABT-888) (RP2D) in combination with cisplatin plus gemcitabine.

III. Document anti-tumor activity of veliparib (ABT-888), cisplatin, and gemcitabine as assessed by RECIST 1.1.

IV. Determine the plasma pharmacokinetics of veliparib (ABT-888), cisplatin, and gemcitabine.

V. Determine the abundance of gemcitabine triphosphate in PBMCs following gemcitabine administration.

VI. Measure the abundance of DNA-platinum adducts in tumor tissue following cisplatin administration.

VII. Measure PARP enzymatic activity in PBMC and tumor tissue following study treatment.

VIII. Perform an exploratory correlation between abundance of BRCA and other proteins assessed by tumor immunohistochemistry and clinical response.

OUTLINE: This is a multicenter, dose-escalation study of veliparib and gemcitabine hydrochloride. Patients are stratified according to presence of suspected or known BRCA mutations (no vs yes).

Patients receive veliparib orally every 12 hours on days 1-12, gemcitabine hydrochloride IV over 30 minutes on days 3 and 10, and cisplatin IV over 60-120 minutes on day 3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with suspected or known germline BRCA mutations may continue to receive single-agent veliparib continuously in the absence of disease progression or unacceptable toxicity. Patients may undergo blood, tumor tissue, and hair follicle sample collection periodically for pharmacokinetic and correlative studies.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed advanced biliary/pancreatic cancer, urothelial cancer, or non-small cell lung cancer that is metastatic or unresectable
* Patients with known CNS metastases should be excluded from this clinical trial
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%)
* Life expectancy of greater than 12 weeks
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin within normal institutional limits
* AST/ALT ≤ 2.5 times institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance ≥ 60 mL/min
* QTc interval on ECG ≤ 0.48 seconds by Bazett's calculation (≤ CTCAE v.4 grade 2)
* Not pregnant or nursing
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Patients must be able to swallow pills and have no significant impairment in gastrointestinal absorption
* Patients with known or suspected germline mutation in BRCA1 or BRCA2 are eligible to participate

  * Patients in study screening (primarily those with pancreatic cancer) who have a family history that is suspicious for BRCA1 or BRCA2 germline mutation should be assessed by the BRCAPRO computer program to quantitate the likelihood of harboring a deleterious BRCA mutation
  * Patients found to have a BRCAPRO probability score of ≥ 20% should undergo formal full-sequence BRCA testing
  * Patients in screening with a BRCAPRO probability of ≥ 20% who decline genetic testing are not eligible to participate in this trial due to the potential to confound safety assessment
* No uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* HIV-positive patients are eligible
* No active seizure or history of seizure disorder
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to veliparib (ABT-888) or other agents used in this study
* No peripheral neuropathy greater than grade1
* No prior systemic treatment
* No prior cytotoxic chemotherapy (neoadjuvant, adjuvant, or metastatic setting)
* At least 4 weeks since major surgery or radiation therapy
* Patients may not be receiving any other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose of veliparib in combination with cisplatin and gemcitabine | 21 days
  The maximum toxicity for each category of interest that are determined to be possibly, probably or definitely related to study treatment will be recorded for each patient and the summary results will be tabulated (according to CTCAE v4.0).

SECONDARY OUTCOMES:
Dose-limiting and other toxicities according to CTCAE v4.0 | Up to 4 weeks post-treatment
Recommended phase II dose | Up to 4 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Appleman, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania